CLINICAL TRIAL: NCT01597401
Title: A Phase 1, Placebo-Controlled, Randomized, Double-Blind Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Escalating, Single Oral Doses of Aes-103 in Subjects With Stable Sickle Cell Disease
Brief Title: A Single Dose Study of the Safety, Blood Levels and Biological Effects of Aes-103 Compared to Placebo in Subjects With Stable Sickle Cell Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Collaborators: SAIC-Frederick, Inc. (Industry); Therapeutics for Rare and Neglected Diseases (TRND) (NIH); QS Pharma (Unknown); National Chung Cheng University (Other); Infrared Imaging and Thermometry Unit, Biomedical Engineering and Physical Science Shared Resource (NIBIB) (Unknown); ClinPharm Consulting, LLC (Unknown); Ricerca Biosciences LLC (Unknown); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Cato Research (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Aes-103-002; 1ZIAHL006149-01 (NIH)
Record Dates: First submitted 2012-04-26; First posted 2012-05-14 (Estimated); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Sickle Cell Disease
Keywords: Antisickling Agents
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — 5-hydroxymethylfurfural

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Aes-103 300 mg to 1000 mg (Group A) (Experimental): Group A will consist of six subjects receiving a single dose of either a low dose of Aes-103 (300 mg) or placebo without food. After a minimum of a 1- to 2-week washout period and evaluation of blinded safety data, subjects initially randomized to Aes-103 will receive a second, higher dose of Aes-103 (1,000 mg), and subjects initially randomized to placebo will receive a second dose of placebo without food.
  Interventions: Drug: Aes-103; Drug: Placebo
- Aes-103 2000 mg to 4000 mg (Group B) (Experimental): Group B will consist of six subjects receiving an initial dose of either Aes 103 (2,000 mg) or placebo without food. After a minimum of a 1- to 2-week washout period and evaluation of blinded safety data, subjects initially randomized to Aes-103 will receive a second, higher dose of Aes-103 (4,000 mg), and subjects initially randomized to placebo will receive a second dose of placebo without food.
  Interventions: Drug: Aes-103; Drug: Placebo
- Top Dose Expansion (Group C) (Experimental): Once the top dose (i.e., highest tolerated) of Aes-103 has been determined, the size of this group will be expanded with an additional six subjects (Group C) for a total of 12 at that dose, distributed so that six subjects receiving hydroxyurea (HU) and six subjects not receiving HU (for the past 6 months) will receive study drug (five receiving Aes-103 and one receiving placebo in each of the HU and non-HU treated cohorts). This total of 12 subjects includes the initial six subjects who received the highest dose in the study plus six Group C subjects. These subjects will receive a single dose of the top dose of Aes-103 or placebo without food. After a minimum of a 1- to 2-week washout period and evaluation of blinded safety data, subjects initially randomized to Aes-103 will receive a second dose of the top dose of Aes-103 and subjects initially randomized to placebo will receive a second dose of placebo; all subjects will be administered a pre-dose, high fat, high protein meal.
  Interventions: Drug: Aes-103; Drug: Placebo

INTERVENTIONS:
Drug: Aes-103 — 300 mg Aes-103 powder reconstituted in orange juice to a volume of 100 mL per single dose for oral administration.
  Arms: Aes-103 300 mg to 1000 mg (Group A)
Drug: Aes-103 — 1000 mg Aes-103 powder reconstituted in orange juice to a volume of 100 mL per single dose for oral administration.
  Arms: Aes-103 300 mg to 1000 mg (Group A)
Drug: Aes-103 — 2000 mg Aes-103 powder reconstituted in orange juice to a volume of 100 mL per single dose for oral administration.
  Arms: Aes-103 2000 mg to 4000 mg (Group B)
Drug: Aes-103 — 4000 mg Aes-103 powder reconstituted in orange juice to a volume of 100 mL per single dose for oral administration.
  Arms: Aes-103 2000 mg to 4000 mg (Group B); Top Dose Expansion (Group C)
Drug: Placebo — Orange juice vehicle, a solution that is highly similar in appearance to the Aes-103 orange juice solution.

SUMMARY:
The purpose of this study is to assess the safety, tolerability, pharmacokinetic, and pharmacodynamic effects of Aes-103 (active ingredient 5-hydroxymethyl-2-furfural [5-HMF]) compared with placebo in subjects with stable sickle cell disease (SCD). Safety will be measured by monitoring adverse events (AEs), electrocardiograms (ECGs), vital signs, and laboratory values. Pharmacokinetics of Aes-103 will be measured over time in plasma, red blood cell hemolysate and binding of Aes-103 to hemoglobin. Pharmacodynamic effects will be assessed by measuring partial pressure of oxygen at which 50% of hemoglobin is saturated with oxygen (p50) while breathing normal air, blood oxygen levels (SpO2), ex-vivo antisickling effects in a hypoxic environment, and by imaging related changes in tissue blood flow and oxygen levels.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female, aged 18-65 years old, inclusive
* Have sickle cell disease (SCD) (hemoglobin SS) without hospitalization for pain crises in the 30 days before screening or for any SCD complications on more than two occasions in the past 12 months; subjects are allowed concomitant usage of hydroxyurea (HU) if the dosage is stable for the 2 months before screening and is at a dosage that does not exceed the product's labeling.
* Have normal laboratory values as defined below:

  * Direct bilirubin 0.1 to 1.0 mg/dL
  * Alanine transaminase (serum glutamic pyruvic transaminase) 6 to 41 IU/L
  * Creatinine for females 0.56 to 1.16 mg/dL and for males 0.77 to 1.19 mg/dL
* If female, be non-pregnant and non-breastfeeding and be surgically sterile or using an acceptable method of contraception throughout the study and for 30 days after study completion
* Have successfully completed an outpatient screening visit consisting of medical history, physical examination, 12-lead ECG, vital signs, hematology and chemistry tests, urinalysis, urine drug screen, pregnancy test (females), hemoglobin electrophoresis, hepatitis B and C screening, and HIV serology (Note: Subjects with abnormal screening values may be eligible if the results are not clinically significant, as judged by the investigator or medical monitor)
* Be able to understand and have provided written informed consent including signature on an informed consent form approved by an institutional review board
* Agree to abide by the study schedule and dietary restrictions and to return for the required assessments
* Be willing to abstain from foods high in 5-HMF (e.g., coffee, malt, barley, balsamic vinegar, dried fruits, and caramel products) for at least 3 days before each dosing

Exclusion Criteria:

* Have evidence of clinically significant cardiovascular, respiratory, renal, hepatic, pulmonary, gastrointestinal, hematological, neurological, psychiatric, or other disease that may interfere with the objectives of the study or the safety of the subject, as judged by the investigator in agreement with the sponsor or medical monitor, or have been hospitalized in the past 6 months as a result of these conditions
* Have been hospitalized in the 14 days before enrollment, for any reason
* Be currently on regularly scheduled transfusions
* Have received a transfusion within 2 weeks of administration of study drug
* Have taken herbal preparations in the 2 weeks before dosing (Note: subjects are allowed concomitant usage of HU and other scheduled prescription drugs if the dosage is stable for the 2 months before screening and is at a dosage that does not exceed the product's labeling. These scheduled prescription medications will be continued during the study [including during dosing]. All other medications, including over-the-counter medications used according to the product labeling, administered on an as-needed basis will be permitted except for the 24 hour period before dosing and the day of dosing. Medications for pain management will be allowed as needed [including during dosing.])
* Have taken any other investigational drug within 30 days or 5 half-lives before the screening visit, whichever is longer
* Consumed more than 14 alcoholic drinks per week or more than 3 drinks per day at any point in the past month
* Have received disulfiram or 4-methylpyrazole within 30 days before dosing
* Have taken any cough-cold product containing dextrorphan or dextromethorphan within 4 days before dosing
* Have positive result for urine drug test (cocaine, marijuana, opiates, amphetamines, methamphetamines, benzodiazepines, ethanol) at screening visit. However, use of opiates, amphetamines, or benzodiazepines is allowed if prescribed by a physician.
* Have engaged in strenuous exercise within 72 hours prior to dosing
* Be considered not suitable for participation in this study for any reason, as judged by the investigator
* Have pre-existing allergic or other adverse reactions to orange juice

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-05-12 (Actual); Primary Completion 2013-06-07 (Actual); Study Completion 2013-06-07 (Actual)

PRIMARY OUTCOMES:
Safety, as assessed by frequency and severity of adverse events (AEs), and changes in vital signs, 12-lead electrocardiograms (ECGs), and laboratory assessments as compared to baseline. | 32 days

SECONDARY OUTCOMES:
Plasma area under the curve (AUC) of Aes-103 | predose, .1 hrs, .25 hrs, .5 hrs, .75 hrs, 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr, and 24 hr
Red blood cell (RBC) hemolysate AUC of Aes-103 | predose, .1 hrs, .25 hrs, .5 hrs, .75 hrs, 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr, and 24 hr
Hemoglobin bound 5-hydroxymethyl-2-furfural (5-HMF) AUC | predose, .5 hrs, 1 hr, 4 hr, and 12 hr
Renal elimination of Aes-103 | predose, 0-4hrs, 4-8hrs, and 8-24hrs
Percentage of hemoglobin bound to Aes-103 | predose, 1 hr, 2 hr, 4 hr, and 12 hr
Change from baseline in resting oxygen saturation (SpO2) | predose, .5 hrs, 1 hr, 4 hr, and 12 hr
Change from baseline in partial pressure of oxygen required to achieve 50% hemoglobin saturation (p50) value | predose, 1 hr, 2 hr, 4 hr, and 12 hr
Effects of food ingested prior to dosing on plasma AUC of Aes-103 | predose, .1 hrs, .25 hrs, .5 hrs, .75 hrs, 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr, and 24 hr
Percentage of sickled cells under normal ex vivo conditions | predose, 1 hr, 2 hr, 4 hr, and 12 hr
Change from baseline in blood flow distribution | predose and .5 to 2 hr
Change from baseline in peripheral arterial tonometry | predose and .5 to 2 hr
Change from baseline in pain as measured by the Numerical Pain Rating Scale (NPRS) | -1hr, -.5hrs, -5min, .1hrs, .25 hrs, .5 hrs, .75 hrs, 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr, and 24 hr
Plasma maximum concentration (Cmax) of Aes-103 | predose, .1 hrs, .25 hrs, .5 hrs, .75 hrs, 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr, and 24 hr
Plasma time to maximum concentration (Tmax) of Aes-103 | predose, .1 hrs, .25 hrs, .5 hrs, .75 hrs, 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr, and 24 hr
Plasma half life (t1/2) of Aes-103 | predose, .1 hrs, .25 hrs, .5 hrs, .75 hrs, 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr, and 24 hr
Plasma AUC of Aes-103's metabolite, 5-hydroxymethyl-2-furoic acid (HMFA) | predose, .1 hrs, .25 hrs, .5 hrs, .75 hrs, 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr, and 24 hr
Plasma maximum concentration (Cmax) of HMFA | predose, .1 hrs, .25 hrs, .5 hrs, .75 hrs, 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr, and 24 hr
Plasma time to maximum concentration (Tmax) of HMFA | predose, .1 hrs, .25 hrs, .5 hrs, .75 hrs, 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr, and 24 hr
Plasma half life (t1/2) of HMFA | predose, .1 hrs, .25 hrs, .5 hrs, .75 hrs, 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr, and 24 hr
RBC hemolysate Cmax of Aes-103 | predose, .1 hrs, .25 hrs, .5 hrs, .75 hrs, 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr, and 24 hr
RBC hemolysate Tmax of Aes-103 | predose, .1 hrs, .25 hrs, .5 hrs, .75 hrs, 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr, and 24 hr
RBC hemolysate t1/2 of Aes-103 | predose, .1 hrs, .25 hrs, .5 hrs, .75 hrs, 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr, and 24 hr
RBC hemolysate AUC of HMFA | predose, .1 hrs, .25 hrs, .5 hrs, .75 hrs, 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr, and 24 hr
RBC hemolysate Cmax of HMFA | predose, .1 hrs, .25 hrs, .5 hrs, .75 hrs, 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr, and 24 hr
RBC hemolysate Tmax of HMFA | predose, .1 hrs, .25 hrs, .5 hrs, .75 hrs, 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr, and 24 hr
RBC hemolysate t1/2 of HMFA | predose, .1 hrs, .25 hrs, .5 hrs, .75 hrs, 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr, and 24 hr
Hemoglobin bound 5-HMF Cmax | predose, .5 hrs, 1 hr, 4 hr, and 12 hr
Hemoglobin bound 5-HMF Tmax | predose, .5 hrs, 1 hr, 4 hr, and 12 hr
Hemoglobin bound 5-HMF t1/2 | predose, .5 hrs, 1 hr, 4 hr, and 12 hr
Renal elimination of HMFA | predose, 0-4hrs, 4-8hrs, and 8-24hrs
Effects of food ingested prior to dosing on plasma Cmax of Aes-103 | predose, .1 hrs, .25 hrs, .5 hrs, .75 hrs, 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr, and 24 hr
Effects of food ingested prior to dosing on plasma Tmax of Aes-103 | predose, .1 hrs, .25 hrs, .5 hrs, .75 hrs, 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr, and 24 hr
Effects of food ingested prior to dosing on plasma t1/2 of Aes-103 | predose, .1 hrs, .25 hrs, .5 hrs, .75 hrs, 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr, and 24 hr
Percentage of sickled cells under hypoxic ex vivo conditions | predose, 1 hr, 2 hr, 4 hr, and 12 hr
Change from baseline in vasomotion | predose and .5 to 2 hr

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- US National Institutes of Health - National Heart, Lung, and Blood Institute, Bethesda, Maryland, United States

REFERENCES:
- [Background] Abdulmalik O, Safo MK, Chen Q, Yang J, Brugnara C, Ohene-Frempong K, Abraham DJ, Asakura T. 5-hydroxymethyl-2-furfural modifies intracellular sickle haemoglobin and inhibits sickling of red blood cells. Br J Haematol. 2005 Feb;128(4):552-61. doi: 10.1111/j.1365-2141.2004.05332.x. PMID 15686467
- [Background] Buchanan G, Vichinsky E, Krishnamurti L, Shenoy S. Severe sickle cell disease--pathophysiology and therapy. Biol Blood Marrow Transplant. 2010 Jan;16(1 Suppl):S64-7. doi: 10.1016/j.bbmt.2009.10.001. Epub 2009 Oct 9. PMID 19819341
- [Background] Czok G. [Tolerance of 5-hydroxymethylfurfural (HMF). 2d communication: pharmacologic effects]. Z Ernahrungswiss. 1970 Dec;10(2):103-10. doi: 10.1007/BF02021840. No abstract available. German. PMID 5492127
- [Background] Germond JE, Philippossian G, Richli U, Bracco I, Arnaud MJ. Rapid and complete urinary elimination of [14C]-5-hydroxymethyl-2-furaldehyde administered orally or intravenously to rats. J Toxicol Environ Health. 1987;22(1):79-89. doi: 10.1080/15287398709531052. PMID 3612837
- [Background] Godfrey VB, Chen LJ, Griffin RJ, Lebetkin EH, Burka LT. Distribution and metabolism of (5-hydroxymethyl)furfural in male F344 rats and B6C3F1 mice after oral administration. J Toxicol Environ Health A. 1999 Jun 11;57(3):199-210. doi: 10.1080/009841099157764. PMID 10376886
- [Background] Lo Coco F, Novelli V, Valentini C, Ceccon L. High-performance liquid chromatographic determination of 2-furaldehyde and 5-hydroxymethyl-2-furaldehyde in fruit juices. J Chromatogr Sci. 1997 Dec;35(12):578-83. doi: 10.1093/chromsci/35.12.578. PMID 9397542
- [Background] Matzi V, Lindenmann J, Muench A, Greilberger J, Juan H, Wintersteiger R, Maier A, Smolle-Juettner FM. The impact of preoperative micronutrient supplementation in lung surgery. A prospective randomized trial of oral supplementation of combined alpha-ketoglutaric acid and 5-hydroxymethylfurfural. Eur J Cardiothorac Surg. 2007 Nov;32(5):776-82. doi: 10.1016/j.ejcts.2007.07.016. Epub 2007 Sep 4. PMID 17768058
- [Background] Mitchell BL. Sickle cell trait and sudden death--bringing it home. J Natl Med Assoc. 2007 Mar;99(3):300-5. PMID 17393956
- [Background] Mrochek JE, Rainey WT Jr. Identification and biochemical significance of substituted furans in human urine. Clin Chem. 1972 Aug;18(8):821-8. No abstract available. PMID 5043270
- [Background] Murkovic M, Pichler N. Analysis of 5-hydroxymethylfurfual in coffee, dried fruits and urine. Mol Nutr Food Res. 2006 Sep;50(9):842-6. doi: 10.1002/mnfr.200500262. PMID 16917810
- [Background] Platt OS. Hydroxyurea for the treatment of sickle cell anemia. N Engl J Med. 2008 Mar 27;358(13):1362-9. doi: 10.1056/NEJMct0708272. No abstract available. PMID 18367739
- [Background] Prior RL, Wu X, Gu L. Identification and urinary excretion of metabolites of 5-(hydroxymethyl)-2-furfural in human subjects following consumption of dried plums or dried plum juice. J Agric Food Chem. 2006 May 17;54(10):3744-9. doi: 10.1021/jf0601113. PMID 19127754
- [Background] Simonian TA. [Toxico-hygienic characteristics of oxymethylfurfural]. Vopr Pitan. 1969 Jan-Feb;28(1):54-8. No abstract available. Russian. PMID 4312377
- [Background] Zakhari S. Overview: how is alcohol metabolized by the body? Alcohol Res Health. 2006;29(4):245-54. PMID 17718403